CLINICAL TRIAL: NCT01670656
Title: A Multicenter, Randomized, Partially Blinded, Placebo-controlled Clinical Trial to Evaluate the Effect on Primary Dysmenorrhea of Vaginal Rings With an Average Daily Release of 700 μg Nomegestrol Acetate (NOMAC) and 300 μg Estradiol (E2), or 900 μg Nomegestrol Acetate (NOMAC) and 300 μg Estradiol (E2), or 100 μg Etonogestrel (ENG) and 300 μg E2, or 125 μg Etonogestrel (ENG) and 300 μg E2. Protocol MK-8175A/MK-8342B 057 (Abbreviated as P057), Also Known as SCH900121/SCH900432 08257 (Abbreviated as P08257)
Brief Title: A Study to Evaluate the Effect of Contraceptive Vaginal Rings on Primary Dysmenorrhea (P08257/MK-8175A/MK-8342B-057)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08257; 2012-002449-40 (EudraCT Number); MK-8175A/MK-8342B-057 (Other: Merck)
Record Dates: First submitted 2012-08-14; First posted 2012-08-22 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- NOMAC-E2 700/300 mcg (Experimental): NOMAC-E2 700/300 mcg will be administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Nomegestrol acetate contraceptive vaginal ring (NOMAC-CVR); Drug: Ibuprofen
- NOMAC-E2 900/300 mcg (Experimental): NOMAC-E2 900/300 mcg will be administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Nomegestrol acetate contraceptive vaginal ring (NOMAC-CVR); Drug: Ibuprofen
- ENG-E2 100/300 mcg (Experimental): ENG-E2 100/300 mcg will be administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Etonogestrel containing contraceptive vaginal ring (ENG-CVR); Drug: Ibuprofen
- ENG-E2 125/300 mcg (Experimental): ENG-E2 125/300 mcg will be administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Etonogestrel containing contraceptive vaginal ring (ENG-CVR); Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo will be administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Placebo; Drug: Ibuprofen

INTERVENTIONS:
Drug: Nomegestrol acetate contraceptive vaginal ring (NOMAC-CVR) — Either 700 or 900 mcg NOMAC and 300 mcg E2 intravaginal ring for two 28-day cycles
  Other Names: SCH900121; MK-8175A
  Arms: NOMAC-E2 700/300 mcg; NOMAC-E2 900/300 mcg
Drug: Etonogestrel containing contraceptive vaginal ring (ENG-CVR) — Either 100 or 125 mcg ENG and 300 mcg E2, intravaginally for two 28-day cycles
  Other Names: SCH900432; MK-8342B
  Arms: ENG-E2 100/300 mcg; ENG-E2 125/300 mcg
Drug: Placebo — Placebo to match vaginal ring, intravaginally for two 28-day cycles
  Arms: Placebo
Drug: Ibuprofen — Ibuprofen 400 mg will be dispensed throughout the entire study as needed as rescue medication for treating menstrual cramping pain. The maximum daily ibuprofen dose is 3200 mg (8 tablets)
  Other Names: Motrin

SUMMARY:
The study investigates four vaginal ring groups with respect to relief of primary dysmenorrhea, and should identify at least one vaginal ring that shows clinically relevant treatment efficacy in relief of primary dysmenorrhea.

DETAILED DESCRIPTION:
The study investigates four vaginal ring groups with respect to relief of primary dysmenorrhea, and should identify at least one vaginal ring that shows clinically relevant treatment efficacy in relief of primary dysmenorrhea. The intake of ibuprofen rescue medication and the impact on daily life is investigated: change from baseline data of these two variables will be compared between each of the four active ring groups, separately, and the placebo ring group. Furthermore, the study assesses the measurement characteristics and psychometric properties of a newly developed Dysmenorrhea Daily Dairy. Vaginal bleeding pattern and general safety and tolerability will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 and ≤35
* Established diagnosis of primary dysmenorrhea
* If of child-bearing potential must agree to use condoms for contraception during the entire screening period, treatment period, and post-treatment period until the final study visit, unless she or her partner are surgically sterilized
* Agree to stop using hormonal contraceptive (combined or progestin-only), or a non hormonal intrauterine device (IUD)
* Regular menstrual cycles ranging from 24 to 35 days in length

Exclusion Criteria:

* Any of the following contraindications to the use of contraceptive steroids including: presence or a history of venous or arterial thrombotic/thromboembolic events or cerebrovascular accident (stroke, history of migraine with focal neurological symptoms, diabetes mellitus with vascular involvement, severe or multiple risk factor(s) for venous or arterial thrombosis, severe dyslipoproteinemia, severe hypertension, pancreatitis or a history thereof if associated with severe hypertriglyceridaemia, presence or history of severe hepatic (liver) disease, including benign or malignant tumors, known or suspected sex steroid-influenced malignancies, and/or undiagnosed vaginal bleeding
* Pregnant or breastfeeding
* Secondary dysmenorrhea
* Has not had spontaneous menstruation following a delivery or abortion
* Participated in an investigational drug study within 30 days
* History of malignancy ≤5 years
* Documented abnormal cervical smear result within 6 months
* Use of recreational or illicit drugs
* Consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking
* Allergy/sensitivity to ibuprofen, or any contraindication to its use, or has experienced asthma, urticaria, or allergic-type reactions after taking aspirin, or other nonsteroidal anti inflammatory drugs
* Has been sterilized using a fallopian tube occlusion device
* Is receiving, or has received sex hormones for any purpose other than contraception within 2 months or injectable hormonal contraception within 6 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 439 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2013-09-11 (Actual); Study Completion 2013-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox MC, Klipping C, Nguyen AM, Frenkl TL, Cruz SM, Wang Y, Korver T. A phase 2b multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of vaginal rings containing nomegestrol acetate or etonogestrel and 17beta-estradiol in the treatment of women with primary dysmenorrhea. Contraception. 2019 Feb;99(2):125-130. doi: 10.1016/j.contraception.2018.10.009. Epub 2018 Nov 12. PMID 30439359

RESULTS

PARTICIPANT FLOW:
Groups:
- NOMAC-E2 700/300 mcg: NOMAC-E2 700/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- NOMAC-E2 900/300 mcg: NOMAC-E2 900/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- ENG-E2 100/300 mcg: ENG-E2 100/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- ENG-E2 125/300 mcg: ENG-E2 125/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Placebo: Placebo was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
Period: Overall Study
Arm/Group | NOMAC-E2 700/300 mcg | NOMAC-E2 900/300 mcg | ENG-E2 100/300 mcg | ENG-E2 125/300 mcg | Placebo
Started | 86 | 91 | 87 | 85 | 90
Treated | 86 | 91 | 86 | 85 | 90
Completed | 83 | 84 | 79 | 79 | 79
Not Completed | 3 | 7 | 8 | 6 | 11
Not completed — Non-compliance with study drug | 0 | 0 | 3 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Non-compliance with protocol | 0 | 3 | 1 | 1 | 2
Not completed — Adverse Event | 2 | 2 | 2 | 3 | 3
Not completed — Subject withdrew consent | 0 | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3
Not completed — Subject moved | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- NOMAC-E2 900/300 mcg: NOMAC-E2 900/300 mcg administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 700/300 mcg | NOMAC-E2 900/300 mcg | ENG-E2 100/300 mcg | ENG-E2 125/300 mcg | Placebo | Total
Number analyzed (Participants) | 86 | 91 | 87 | 85 | 90 | 439
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (7.5) | 28.7 (8.1) | 29.0 (7.7) | 28.3 (7.8) | 28.4 (8.2) | 28.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 91 | 87 | 85 | 90 | 439
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Menstrual Cramping Pain Score Through Cycle 2
Description: The Mean Menstrual Cramping Pain score was calculated as the average of the three highest daily menstrual cramping scores (item #3 of the Menstrual Distress Questionnaire: "Cramps") in the baseline cycle and treatment Cycle 2, respectively. The daily menstrual cramping pain score was based on five pain categories: none (0); mild (1); moderate (2); strong (3); and severe (4). In case of absence of withdrawal bleeding, or onset of menstruation, the mean of the three highest menstrual cramping pain scores recorded within Days 21-28 was used for analysis. The Mean Menstrual Cramping Pain Score in the baseline or subsequent cycles could range from 0 (none) to 4 (severe).
Time Frame: Baseline and Day 29 to 56 (Cycle 2)
Population: All randomized participants in whom a vaginal ring was inserted and who had at least one baseline or one post-baseline value for Menstrual Cramping Pain Score
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | NOMAC-E2 700/300 mcg | NOMAC-E2 900/300 mcg | ENG-E2 100/300 mcg | ENG-E2 125/300 mcg | Placebo
Number analyzed (Participants) | 85 | 91 | 86 | 85 | 90
Units on a scale | -1.7 [-2.0 to -1.5] | -1.7 [-1.9 to -1.5] | -1.9 [-2.1 to -1.7] | -1.7 [-1.9 to -1.5] | -1.2 [-1.4 to -0.9]
Statistical Analysis 1: Comparison: NOMAC-E2 700/300 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -0.6, 95% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 2: Comparison: NOMAC-E2 900/300 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -0.6, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 3: Comparison: ENG-E2 100/300 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -0.8, 95% CI 2-sided [-1.1 to -0.4]
Statistical Analysis 4: Comparison: ENG-E2 125/300 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -0.5, 95% CI 2-sided [-0.9 to -0.2]

2. Secondary Outcome: Change From Baseline in Total Mean Impact Score Through Cycle 2
Description: Total Mean Impact Score is the mean of the sum of the daily responses to questions 6, 8, 9, and 10 in the Dysmenorrhea Daily e-Dairy, as recorded within the menstrual cramping pain analysis window. These questions assessed how much interference there was from pelvic cramping pain on work/school activities (Q6), physical activities (Q8), social/leisure activities (Q9) and sleep (Q10). Each question was rated on a 5-point (0-4) scale, with 0 being "not at all", 1 "slightly", 2 "moderately", 3 "quite a bit" and 4 "extremely". The total mean impact score could thus range from 0 (lowest possible impact) to 16 (highest possible impact).
Time Frame: Baseline and Day 29 to 56 (Cycle 2)
Population: All randomized participants in whom a vaginal ring was inserted and who had at least one baseline or one post-baseline value for Total Mean Impact Score
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | NOMAC-E2 700/300 mcg | NOMAC-E2 900/300 mcg | ENG-E2 100/300 mcg | ENG-E2 125/300 mcg | Placebo
Number analyzed (Participants) | 85 | 90 | 86 | 85 | 90
Units on a scale | -4.8 [-5.6 to -4.0] | -5.0 [-5.7 to -4.2] | -4.7 [-5.5 to -3.9] | -4.3 [-5.1 to -3.5] | -3.1 [-3.9 to -2.4]
Statistical Analysis 1: Comparison: NOMAC-E2 700/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.002, cLDA; Difference in Least Squares Means = -1.7, 95% CI 2-sided [-3.0 to -0.4]
Statistical Analysis 2: Comparison: NOMAC-E2 900/300 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -1.9, 95% CI 2-sided [-3.1 to -0.6]
Statistical Analysis 3: Comparison: ENG-E2 100/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.003, cLDA; Difference in Least Squares Means = -1.6, 95% CI 2-sided [-2.9 to -0.3]
Statistical Analysis 4: Comparison: ENG-E2 125/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.024, cLDA; Difference in Least Squares Means = -1.2, 95% CI 2-sided [-2.5 to 0.1]

3. Secondary Outcome: Change From Baseline in Number of Ibuprofen Tablets Taken Through Cycle 2
Description: Participants were provided with ibuprofen 400 mg tablets at the screening visit to be taken throughout the study as needed as rescue medication for treating menstrual cramping pain. The maximum daily ibuprofen dose was 3200 mg (8 tablets). Participants were instructed to take the provided ibuprofen, and no other medications, for the relief of menstrual cramping pain, and to record their ibuprofen usage in their e-Diaries.
Time Frame: Baseline and Day 29 to 56 (Cycle 2)
Population: All randomized participants in whom a vaginal ring was inserted and who had at least one baseline or one post-baseline value for Number of Ibuprofen Tablets Taken
Measure: Least Squares Mean (95% Confidence Interval); unit: Ibuprofen tablets
Arm/Group | NOMAC-E2 700/300 mcg | NOMAC-E2 900/300 mcg | ENG-E2 100/300 mcg | ENG-E2 125/300 mcg | Placebo
Number analyzed (Participants) | 85 | 91 | 86 | 85 | 90
Ibuprofen tablets | -6.4 [-7.5 to -5.3] | -6.3 [-7.4 to -5.2] | -7.1 [-8.2 to -6.0] | -6.0 [-7.1 to -4.9] | -4.8 [-6.0 to -3.7]
Statistical Analysis 1: Comparison: NOMAC-E2 700/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.026, cLDA; Difference in Least Squares Means = -1.6, 95% CI 2-sided [-3.4 to 0.2]
Statistical Analysis 2: Comparison: NOMAC-E2 900/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.036, cLDA; Difference in Least Squares Means = -1.5, 95% CI 2-sided [-3.3 to 0.2]
Statistical Analysis 3: Comparison: ENG-E2 100/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.002, cLDA; Difference in Least Squares Means = -2.3, 95% CI 2-sided [-4.1 to -0.5]
Statistical Analysis 4: Comparison: ENG-E2 125/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.1, cLDA; Diffference in Least Squares Means = -1.2, 95% CI 2-sided [-3.0 to 0.6]

4. Secondary Outcome: Change From Baseline in Number of Days of Ibuprofen Intake Through Cycle 2
Description: as for outcome 3
Time Frame: Baseline and Day 29 to 56 (Cycle 2)
Population: All randomized participants in whom a vaginal ring was inserted and who had at least one baseline or one post-baseline value for Number of Days of Ibuprofen Intake
Measure: Least Squares Mean (95% Confidence Interval); unit: Days of ibuprofen intake
Arm/Group | NOMAC-E2 700/300 mcg | NOMAC-E2 900/300 mcg | ENG-E2 100/300 mcg | ENG-E2 125/300 mcg | Placebo
Number analyzed (Participants) | 85 | 91 | 86 | 85 | 90
Days of ibuprofen intake | -1.3 [-1.5 to -1.0] | -1.7 [-2.0 to -1.4] | -1.7 [-2.0 to -1.4] | -1.4 [-1.7 to -1.1] | -1.1 [-1.4 to -0.9]
Statistical Analysis 1: Comparison: NOMAC-E2 700/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.447, cLDA; Difference in Least Squares Means = -0.1, 95% CI 2-sided [-0.6 to 0.3]
Statistical Analysis 2: Comparison: NOMAC-E2 900/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.003, cLDA; Difference in Least Squares Means = -0.6, 95% CI 2-sided [-1.0 to -0.1]
Statistical Analysis 3: Comparison: ENG-E2 100/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.003, cLDA; Difference in Least Squares Means = -0.6, 95% CI 2-sided [-1.0 to -0.1]
Statistical Analysis 4: Comparison: ENG-E2 125/300 mcg vs Placebo; Test type: Superiority or Other; p = 0.156, cLDA; Difference in Least Squares Means = -0.3, 95% CI 2-sided [-0.7 to 0.2]

ADVERSE EVENTS:
Time Frame: Up to 64 days
Description: The Safety Analysis was based on all randomized participants in whom a vaginal ring was inserted.
Groups:
- NOMAC-E2 (700/300 mcg): NOMAC-E2 700/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days
- NOMAC-E2 (900/300 mcg): NOMAC-E2 900/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- ENG-E2 (100/300 mcg): ENG-E2 100/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- ENG-E2 (125/300 mcg): ENG-E2 125/300 mcg was administered for two 28-day treatment periods, each period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
Arm/Group | NOMAC-E2 (700/300 mcg) | NOMAC-E2 (900/300 mcg) | ENG-E2 (100/300 mcg) | ENG-E2 (125/300 mcg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/91 | 0/86 | 1/85 | 0/90
Other Adverse Events (participants affected / at risk) | 12/86 | 11/91 | 14/86 | 7/85 | 11/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (700/300 mcg) (N=86) | NOMAC-E2 (900/300 mcg) (N=91) | ENG-E2 (100/300 mcg) (N=86) | ENG-E2 (125/300 mcg) (N=85) | Placebo (N=90)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (700/300 mcg) (N=86) | NOMAC-E2 (900/300 mcg) (N=91) | ENG-E2 (100/300 mcg) (N=86) | ENG-E2 (125/300 mcg) (N=85) | Placebo (N=90)
Headache (Nervous system disorders) | 9 (13) | 9 (19) | 11 (13) | 5 (7) | 7 (9)
Breast pain (Reproductive system and breast disorders) | 5 (7) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including slides and texts of oral or other public presentations and texts of any transmission through any electronic media that report results of the trial. The Sponsor has the right to review and comment with respect to publications, abstracts, slides, and manuscripts, as wells as comment on the data analysis and presentation.